CLINICAL TRIAL: NCT05495022
Title: he Effect of MBSR (Conscious Awareness-Based Stress Reduction) Program on Anxiety, Work-Related Emotional Burnout and Job Satisfaction in Midwives
Brief Title: The Effect of MBSR (Mindfulness-Based Stress Reduction) Program on Anxiety, Work-Related Emotional Burnout and Job Satisfaction in Midwives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Sıdıka Özlem CENGİZHAN, : Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 28-02-2022 / 26
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Midwives; Mindfulness; Anxiety; Professional Burnout; Job Satisfaction
MeSH Terms: conditions — Anxiety Disorders; Burnout, Professional | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBSR group (Experimental): Mindfulness-based stress reduction (MBSR) program
  Interventions: Behavioral: Mindfulness-based stress reduction (MBSR) program
- Control group (No Intervention): standard care group

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction (MBSR) program — Mindfulness-based stress reduction (MBSR) program will be applied by the researcher to the midwives in the experimental group. Conscious Awareness-Based Stress Reduction will be applied by the researcher (S.Ö.C.) who has received training (16 hours) and has a certificate in this field. Stress reduction program based on mindfulness is planned as 2 sessions per week for 4 weeks, a total of 8 sessions. Each session is planned to last 40-60 minutes on average. Sessions will continue as individual and group sessions by determining the days when midwives are available online.
  Arms: MBSR group

SUMMARY:
Mindfulness; It is the state of paying attention and being aware of what is happening right now. Mindfulness, includes noticing what is happening in the present moment and the way of meeting all that is noticed.

The research will be conducted in a randomized controlled manner in order to determine the Effect of MBSR (Conscious Awareness Based Stress Reduction) Program on Anxiety, Work Related Emotional Burnout and Job Satisfaction in midwives.

Data will be collected from midwives working at Gaziantep Cengiz Gökçek Gynecology and Childhood Hospital between September 1 and December 30, 2022. Midwives who agree to participate in the study and meet the criteria will be sent and asked to fill in web-based online questionnaires (Whatsapp) prepared by the researchers through Google Forms. As a pre-test, "Descriptive Information Form", "Beck Anxiety Scale (BAI)", "Work-Related Emotional Burnout Scale" and "Minnesota Job Satisfaction Scale (MSQ) Short Form" will be administered to midwives in the experimental and control groups. After the stress reduction program based on mindfulness was applied online by the researcher to the experimental group, 2 sessions a week for 4 weeks (1 month), a total of 8 sessions; Post-test data will be obtained by re-applying the "Beck Anxiety Scale (BAS)", "Work-Related Emotional Burnout Scale" and "Minnesota Job Satisfaction Scale (MSQ) Short Form" scale to the experimental group and simultaneously to the control group.

The universe of the research will be composed of midwives working at Gaziantep Cengiz Gökçek Gynecology and Childhood Hospital on the relevant dates. The minimum number of individuals to be included in the sample of the study was determined by power analysis. Sample size when power analysis is done; Assuming that the method applied with 5% error level, bidirectional significance level, 95% confidence interval and 80% ability to represent the universe, would reduce the anxiety score averages (8.20±8.64) by 6 points, a total of 66 midwives (33 experimental, 33 control) calculated. A total of 80 midwives (40 experimental, 40 control) are planned to be included in the study, taking into account possible case losses (approximately 20%).

DETAILED DESCRIPTION:
Mindfulness; It is the state of paying attention and being aware of what is happening right now. Mindfulness includes noticing what is happening in the present moment and the way of meeting all that is noticed.

The research will be conducted in a randomized controlled manner in order to determine the Effect of MBSR (Conscious Awareness Based Stress Reduction) Program on Anxiety, Work Related Emotional Burnout and Job Satisfaction in midwives.

Data will be collected from midwives working at Gaziantep Cengiz Gökçek Gynecology and Childhood Hospital between September 1 and December 30, 2022. Midwives who agree to participate in the study and meet the criteria will be sent and asked to fill in web-based online questionnaires (Whatsapp) prepared by the researchers through Google Forms. As a pre-test, "Descriptive Information Form", "Beck Anxiety Scale (BAI)", "Work-Related Emotional Burnout Scale" and "Minnesota Job Satisfaction Scale (MSQ) Short Form" will be administered to midwives in the experimental and control groups. After the stress reduction program based on mindfulness was applied online by the researcher to the experimental group, 2 sessions a week for 4 weeks (1 month), a total of 8 sessions; Post-test data will be obtained by re-applying the "Beck Anxiety Scale (BAS)", "Work-Related Emotional Burnout Scale" and "Minnesota Job Satisfaction Scale (MSQ) Short Form" scale to the experimental group and simultaneously to the control group.

The universe of the research will be composed of midwives working at Gaziantep Cengiz Gökçek Gynecology and Childhood Hospital on the relevant dates. The minimum number of individuals to be included in the sample of the study was determined by power analysis. Sample size when power analysis is done; Assuming that the method applied with 5% error level, bidirectional significance level, 95% confidence interval and 80% ability to represent the universe, would reduce the anxiety score averages (8.20±8.64) by 6 points, a total of 66 midwives (33 experimental, 33 control) calculated. A total of 80 midwives (40 experimental, 40 control) are planned to be included in the study, taking into account possible case losses (approximately 20%).

Data Collection Form and Tools Data will be collected with "Descriptive Information Form", "Beck Anxiety Scale (BAI)", "Work-Related Emotional Burnout Scale" and "Minnesota Job Satisfaction Scale (MSQ) Short Form".

Midwifery Initiative Mindfulness-based stress reduction (MBSR) program will be applied by the researcher to the midwives in the experimental group. Conscious Awareness-Based Stress Reduction will be applied by the researcher (S.Ö.C.) who has received training (16 hours) and has a certificate in this field. Stress reduction program based on mindfulness is planned as 2 sessions per week for 4 weeks, a total of 8 sessions. Each session is planned to last 40-60 minutes on average. Sessions will continue as individual and group sessions by determining the days when midwives are available online.Variables of the Study Dependent Variable: the scores of the midwives from the scales Independent Variable: Applied Mindfulness-Based Stress Reduction (MBSR) program Evaluation of Data Number, percentile distribution, arithmetic mean, chi-square test, standard deviation and Cronbach's α reliability coefficient will be used in the statistical evaluation of continuous and categorical data with SPSS 25.0 (Statistical Program in Social Sciences) program. Kolmogorov Smirnov test will be used to determine whether the data show a normal distribution. If the normal distribution is shown, the t-test will be used in dependent and independent groups; Mann Whitney-U test and Wilcoxon tests will be used in non-normally distributed groups. Significance will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Being a midwifery graduate (High school, undergraduate) Working actively at Gaziantep Cengiz Gökçek Gynecology and Pediatrics Hospital Volunteering to participate in the study be over 18 years old

Exclusion Criteria:

* Not wanting to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2022-06-04 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Beck Anxiety Scale | Change in anxiety at 4 weeks
  It is a 4-point Likert type scale, developed by Beck et al.(1988) and validated in Turkish by Ulusoy et al.(1998), and consists of 21 questions aiming to measure the severity of anxiety. The items of the scale are scored between 0-3 and a high total score indicates an increased level of anxiety and a low score between 8-15 points; A score of 16-25 indicates moderate anxiety, and a score of 26-63 indicates a high level of anxiety.

SECONDARY OUTCOMES:
Work-Related Emotional Burnout Scale | Change in work-related emotional burnout at 4 weeks
  Turkish validity and reliability of the 6-statement and one-dimensional Work-Related Emotional Burnout Scale developed by Wharton (1993), Günay (2021). There is no reverse expression in the scale. It is designed on a 5-point Likert scale with 1 = I never feel this way, 5 = I feel this way every day. The higher the sum of statements, the higher the level of burnout.
Minnesota Job Satisfaction Scale (MSQ) Short Form | Change in job satisfaction in 4 weeks
  Minnesota Job Satisfaction Scale is one of the most common indices used to measure job satisfaction of employees. The scale developed by Weiss, Dawis, England, and Lofquist has two forms, the long form and short form. each item is arranged with Likert type scoring and ranging from 1 to 5; It consists of 20 items with the statements "I am not at all satisfied", "I am not satisfied", "I am undecided", "I am satisfied", "I am very satisfied". In the evaluation of the options, the highest score is 100 and the lowest score is 20. A score of 20-39 indicates very low, a score of 40-59 indicates low, a score of 60-79 indicates sufficient, and a score of 80-100 indicates high satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Science, Gaziantep, Şahinbey/ Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mayer B, Polak MG, Remmerswaal D. Mindfulness, Interpretation Bias, and Levels of Anxiety and Depression: Two Mediation Studies. Mindfulness (N Y). 2019;10(1):55-65. doi: 10.1007/s12671-018-0946-8. Epub 2018 Apr 12. PMID 30662572
- [Background] Lin L, He G, Yan J, Gu C, Xie J. The Effects of a Modified Mindfulness-Based Stress Reduction Program for Nurses: A Randomized Controlled Trial. Workplace Health Saf. 2019 Mar;67(3):111-122. doi: 10.1177/2165079918801633. Epub 2018 Oct 29. PMID 30370837
- [Result] Kriakous SA, Elliott KA, Lamers C, Owen R. The Effectiveness of Mindfulness-Based Stress Reduction on the Psychological Functioning of Healthcare Professionals: a Systematic Review. Mindfulness (N Y). 2021;12(1):1-28. doi: 10.1007/s12671-020-01500-9. Epub 2020 Sep 24. PMID 32989406